CLINICAL TRIAL: NCT01719796
Title: Assessment of the Ventilatory Effects of Transverse Abdominal Plan Regional Analgesia Following Abdominal Surgery.
Brief Title: Effect of TAP Block on Ventilatory Function Following Abdominal Surgery
Acronym: KTAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Mathieu RAUX, Associate Professor, Pierre and Marie Curie University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTAP
Record Dates: First submitted 2012-10-24; First posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilateral TAP catheter (Experimental): Ultrasonography guided bilateral TAP catheter insertion.
  Interventions: Procedure: Regional analgesia infusion
- No TAP catheter (No Intervention)

INTERVENTIONS:
Procedure: Regional analgesia infusion
  Arms: Bilateral TAP catheter

SUMMARY:
Abdominal surgery impairs ventilation. Postoperative pain accounts for this impairment. Regional analgesia is known to reduce pain, thus to limit ventilatory impairment. The investigators hypothesized bilateral continuous transverse abdominal plan block would reduce ventilatory impairment following abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* laparotomy

Exclusion Criteria:

* below 18, pregnancy, prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
vital capacity | 72h

SECONDARY OUTCOMES:
maximum forced expiratory flow | 72h
analgesic consumption | 72h
pain | 72h
  resting pain, assessed using VAS
diaphragmatic course | 72h
  using ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu RAUX, MD, PhD, Study Director — Pierre et Marie Curie University, Paris, France
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne